CLINICAL TRIAL: NCT03226262
Title: FFRangio Accuracy vs. Standard FFR
Acronym: FAST-FFR
Status: Completed | Type: Observational
Sponsor: CathWorks Ltd. (Industry)
Collaborators: CRF (Unknown)
Responsible Party: Sponsor
Other Study IDs: CWX-03
Record Dates: First submitted 2017-07-12; First posted 2017-07-21 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: FFRangio — FFRangio is a non-invasive image-based software device that provides physicians with a quantitative analysis of functional significance of the coronary lesion, similar to invasive FFR (Fractional Flow Reserve), and a qualitative three-dimensional model of the demonstrated coronary arteries, during routine PCI procedure. The CathWorks FFRangio software device is able to perform all required processing and calculations, based only on angiography images and hemodynamics information that are acquired during the coronary catheterization procedure.
  The CathWorks FFRangioTM technology does not require any additional use of invasive devices, or any additional vasodilation treatment, as required by other known FFR techniques.

SUMMARY:
This is a prospective, observational, multi-center, single-arm, clinical trial designed to assess the efficacy of FFRangio in measuring FFR obtained from angiography compared to Invasive FFR for diagnosing hemodynamically significant coronary stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, >18 years of age.
* Patients with stable angina or unstable angina or NSTEMI, and in whom invasive FFR is being assessed in a non-culprit stenosis in at least one coronary artery.
* Subject is undergoing invasive FFR with Adenosine, ATP or Papaverine used as hyperemic stimulus.
* Provides written, informed consent (where required)

Exclusion Criteria:

* Contraindication for FFR examination or administration of vasodilators.
* Subject is presenting with acute infarct (STEMI) OR has documented prior STEMI on same side (right/left).
* CTO in target vessel.
* Prior CABG, heart transplant or valve surgery, or prior TAVI/TAVR.
* Known LVEF ≤45%.
* Arteries supplying akinetic or severe hypokinetic territories if already known based on prior imaging.
* TIMI Grade 2 or lower at baseline.
* Target lesion involves Left Main (stenosis >50%).
* PCI with stent in target vessel in past 12 months, or target vessel involves in-stent restenosis.
* Severe, diffuse disease defined as the presence of diffuse, serial gross luminal irregularities present in the majority of the coronary tree.
* Target coronary vessel is supplied by major collaterals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with stable angina, unstable angina or NSTEMI who are referred to coronary angiography and have an invasive FFR measurement with vasodilation in at least one coronary artery. Each subject will undergo both the standard invasive FFR and the investigational FFRangio.
Sampling Method: Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the dichotomously scored FFRangio measured index compared to invasive FFR | 1 hour
  Sensitivity and specificity of the dichotomously scored FFRangio measured index per vessel as compared with invasively-derived FFR; Index ≤ 0.80 is scored "positive" while Index > 0.8 is negative.

SECONDARY OUTCOMES:
Continuously scored FFR (FFRangio and Invasive FFR). | 1 hour
  Regression of FFRangio on continuous FFR, with slope, intercept and the correlation coefficient.
Accuracy, Positive predictive value and negative predictive value per vessel and per lesion | 1 hour
Sensitivity and specificity of the dichotomously scored FFRangio measured index per lesion as measured by the site. | 1 hour
Device Success | 1 hour
  The ratio of produced FFRangio values from all FFRangio measurements that were started.
Usability of FFRangio | 1 hour
  A questionnaire will be completed by the user to assess how easy the system is for use and how intuitive it is.
Comprehensiveness of the FFRangio User Manual in providing adequate instructions | 1 hour
  A questionnaire will be completed to measure if the user understands the main parts of the software instructions after reading the Instructions for use.
Procedure related Adverse and Serious Adverse Events | 1 hour
Device related Adverse and Serious Adverse Events | 1 hour

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - Stanford University, Stanford, California
  - Columbia University Medical Center/NewYork Presbyterian Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
- OLV Ziekenhuis, Aalst, Belgium
- Rigs Hospital CPH, Copenhagen, Denmark
- Israel (3):
  - Shaare Zedek Medical Center, Jerusalem
  - HaSharon Hospital, Petah Tikva
  - Rabin Medical Center, Petah Tikva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fearon WF, Achenbach S, Engstrom T, Assali A, Shlofmitz R, Jeremias A, Fournier S, Kirtane AJ, Kornowski R, Greenberg G, Jubeh R, Kolansky DM, McAndrew T, Dressler O, Maehara A, Matsumura M, Leon MB, De Bruyne B; FAST-FFR Study Investigators. Accuracy of Fractional Flow Reserve Derived From Coronary Angiography. Circulation. 2019 Jan 22;139(4):477-484. doi: 10.1161/CIRCULATIONAHA.118.037350. PMID 30586699